CLINICAL TRIAL: NCT03658499
Title: Evaluating the Clinical Utility and Client Acceptability of Video Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rory Newlands (Other)
Responsible Party: Sponsor-Investigator, Rory Newlands, Associate Director of the THRIVE Center, University of Nevada, Reno
Organization: University of Nevada, Reno (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245130-1
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Domestic Violence
Keywords: intimate partner violence; Domestic Violence; Treatment adjuncts; Dialectical behavior therapy

STUDY DESIGN:
Intervention Model Description: Participants will be divided by strata (court mandated vs. voluntary) and randomly assigned to either the experimental or control condition, after completing the two-day skills group, via a research randomizer (Urbaniak & Plous, 2013), which randomly generates numbers that designate the assignment condition of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Those assigned to the experimental condition will be provided with treatment as usual (the two day skills group) and exposure to the video intervention adjuncts.
  two day skills group plus treatment adjuncts
  Interventions: Behavioral: two day skills group plus treatment adjuncts
- control (Other): Those in the control condition will be provided with treatment as usual (the two day skills group) without access to the video intervention adjuncts.
  two day skills group control group
  Interventions: Behavioral: two day skills group control group

INTERVENTIONS:
Behavioral: two day skills group plus treatment adjuncts — The modified dialectical behavior therapy protocol for victims of intimate partner violence dedicates additional time to address validation of self and others in order to mitigate the impact of punishing social relations, and increase the victims' access to positive reinforcement (Iverson et al., 2009). The modified protocol covers the same four major modules as the original DBT protocol in an abbreviated manner. Participants in this group will be provided with the treatment adjuncts.
  Arms: Experimental
Behavioral: two day skills group control group — The modified dialectical behavior therapy protocol for victims of intimate partner violence dedicates additional time to address validation of self and others in order to mitigate the impact of punishing social relations, and increase the victims' access to positive reinforcement (Iverson et al., 2009). The modified protocol covers the same four major modules as the original DBT protocol in an abbreviated manner. Participants in this group will not be provided with the treatment adjuncts and will serve as the control group
  Arms: control

SUMMARY:
Intimate partner violence (IPV) is a common occurrence in the U.S. Victims of IPV are at an elevated risk of experiencing a variety of physical and mental health consequences, which frequently co-occur and act synergistically, placing victims at a higher risk for revictimization. Experts recommend that interventions for victims of IPV focus on helping victims attain more balanced emotions and behaviors, rather than treating specific nosologies. One transdiagnostic treatment, Dialectical Behavior Therapy (DBT), focused on helping individuals gain more balanced emotions and behaviors, has shown success in treating victims of IPV. However, the DBT for IPV treatment protocol is not without it's limitations. Specifically, clients may need additional exposure to the skills and concepts taught in the treatment. Yet, additional exposure to the skills facilitated though a therapist is difficult to do given the limited budgets for services for victims of IPV and the client provider gap. In order to address the client provider gap, increase exposure to the skills, and to increase skills acquisition and generalization, video intervention adjuncts (VIAs) have been developed to serve as treatment adjuncts for the DBT for IPV skills group.

The objective of the current study is to conduct a randomized control trial examining the treatment utility and participant acceptability of the two-day DBT for IPV skills group plus the VIAs versus treatment as usual (the two-day DBT for IPV skills group without the VIAs). The following hypotheses will be examined: 1) those in the experimental VIA condition will experience treatment gains above and beyond those in the control (treatment as usual) condition; 2) those in the experimental VIA condition will view the VIAs as acceptable; and 3) those in the experimental VIA condition will report a greater frequency of using the skills than those in the control condition.

DETAILED DESCRIPTION:
Dialectical Behavioral Therapy as a treatment for IPV victims. Integrating the literature on efficacious cognitive behavioral treatments for disorders such as anxiety, depression, and other emotion regulation difficulties, Linehan developed the framework for DBT.1 In addition to these traditional CBT change-oriented techniques, which may leave clients feeling blamed for their problems or situation, Linehan incorporated radical acceptance. Radical acceptance emphasizes that self-compassion and acceptance (i.e. accepting how things really are rather than how they 'should' be) are necessary for making meaningful changes. When operating from a DBT framework the therapist's goal is to balance and synthesize acceptance and change-oriented strategies. Individuals who have experienced IPV often struggle to accept their situation (e.g. "But I love him," or "he said he will never do it again… although he said that before") and often receive blame from others for their situation (e.g. "Why wouldn't you just leave?"). Treating victims of IPV using a DBT framework allows victims to learn skills to change their situation in a non-judgmental and validating environment.

In addition to providing victims with a validating environment, DBT aims to foster emotion regulation, enhance interpersonal effectiveness, improve self-validation, and increase distress tolerance. Mindfulness (i.e. present-moment awareness, acceptance, and participation without judgment) is core to these skills and to DBT. 2 Overview of the DBT for IPV Treatment Protocol. The DBT for IPV protocol is delivered in a group setting led by two co-therapists. Handouts adapted from the DBT Skills Training: Handouts and Worksheets are provided to clients in session, and homework is provided to help with the retention of the content.3 The DBT for IPV protocol can be broken down into five overarching themes or concepts: mindfulness, emotion regulation, distress tolerance, interpersonal effectiveness, and validation. These concepts form the foundation of the original 12-week closed model, the open group model and the intensive two-day group.4-6 The open group focuses on one module per session, where as the closed group and the two-day group start by introducing the intervention's two foundational topics: mindfulness and behavioral chains. Each module covers several concepts that link back to these two topics.

These five modules were designed to address the psychological sequelae frequently experienced by victims of IPV, as well as to address the underlying mechanisms driving psychological distress among victims of IPV. In addition to reducing revictimization by addressing mental health problems, the DBT for IPV treatment paradigm provides clients with skills (i.e. interpersonal effectiveness and validation) to improve their relationships and reduce the occurrence of violence in their relationships.

Treatment adjuncts. While DBT has demonstrated success in treating a multiple psychological issues, such as suicidal ideation, substance abuse, anger, emotional dysregulation and distress tolerance, it is a costly and time-intensive intervention.7-11 However, research has shown that treatment adjuncts, such as apps and websites, enhance treatment outcomes for a various psychological disorders.12 Technology disseminated interventions have been shown to effectively reduce symptoms of depression, PTSD and anxiety.13 In their review of mobile apps for the treatment of mental disorder, Ameringen and colleagues (2017) noted that employing technology-based interventions might reduce the need for in-person appointments with clinicians, particularly for clients who encounter geographical, time, or financial barriers.13 Further they concluded that apps improve treatment engagement with clinicians and provide opportunities for clinicians to reinforce skills and concepts they taught their clients in session.13 In addition to using treatment adjuncts to enhance treatment outcomes above and beyond treatment as usual, therapists can use treatment adjuncts such as video intervention adjuncts (VIAs), which deliver intervention content via multimedia, as a means of reducing therapist burden.

Research Design and Rationale The objective of this study is to conduct a randomized control trial (RCT) examining the implementation of VIAs, developed for the purpose of enhancing skills generalization, acquisition, and (ultimately) treatment outcomes for DBT for IPV skills group members. Stratified randomization (controlling for those who are court mandated to treatment) will be used assigned participants to the experimental condition (the two-day skills group + the VIAs) or a control condition (the two-day skills group only). The primary outcomes are as follows: 1) investigate whether exposure to the VIA enhances treatment gains above and beyond treatment as usual; 2) assess participant acceptability of the VIAs; and 3) determine if participants in the experimental VIA condition will report a higher frequency of using the skills over the follow-up period than those in the control condition. Following the guidelines for developing and researching behavioral therapies, a Stage One Pilot Trial will be conducted, focusing on feasibility, participant acceptability, and treatment outcome.14 Participants. Following the Onken, Carroll, Shoham, Cuthbert, and Riddle (2014) guidelines for conducting clinical research, a Stage One Pilot Trial will be conducted.15 Stage 1-A is modification or refinement of an existing intervention, and Stage 1-B is feasibility and pilot testing. In this study, the existing intervention is the DBT for IPV skills workshop and the modification is the addition of the VIAs. Because Stage One trials recommend 15-30 subjects per group, the study will require a sample N of 81 (assuming an attrition rate of 35% as reported in Lee and Fruzzetti's 2017 study) to meet the goal N of 60.

Screening and recruitment. Participants will include those who seek services through the THRIVE Center. Community recruitment efforts will include advertising and contacting connections at local community agencies and resource centers for victims of IPV (e.g. temporary protection order offices, Reno Police Department, District Attorney offices, etc.). Individuals interested in receiving treatment will complete intake measures prior to beginning treatment to establish a baseline, at a one-month follow-up, and three-month follow-up.

Intervention. The DBT for IPV skills protocol consists of five major interconnected topics: mindfulness, emotion regulation, distress tolerance, validation, and interpersonal effectiveness. The two-day skills group will be conducted on weekends to increase the likelihood that participants will be able to attend. The skills group will be scheduled from 9am-4pm with a one-hour lunch break (lunch will be provided).

Experimental condition. Participants assigned to the experimental condition will receive a text or email message approximately every two days with a link to a VIA hosted on the online research platform Qualtrics. Each VIA reviews one of the core skills that was taught as part of the two-day skills group. Participants will be asked questions regarding whether the VIA helped them better understand the concept/skill, whether they enjoyed the VIA, and three questions about the content (to serve as a manipulation check). A correct repose to two of the three manipulation check questions will qualify the individual as having completed that VIA.

Control Condition. Participants assigned to the control condition will receive the two-day skills group without the VIAs.

ELIGIBILITY:
Inclusion Criteria:

* Victim of domestic violence
* Must be 18 years old or older
* Speak English
* Have a 8th grade reading level
* Be a female
* Have access to the internet

Exclusion Criteria:

* People who are suicidal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in the difficulties in emotion regulation scale | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  The difficulties in emotion regulation scale is a 36 item self report questionnaire intended to assess multiple aspects of emotion dysregulation. Participants answer on a 1-5 likert scale, with higher scores indicating more problems with emotion regulation. Minimum score = 36 and maximum score = 180. There are six sub scales: Non-acceptance (minimum score = 6 maximum score = 36); difficulties engaging in goal directed behaviors (minimum score = 5 maximum score = 25); impulse control (minimum score = 6 maximum score = 36); lack of emotional awareness (minimum score = 6 maximum score = 36); limited access to emotion regulation strategies (minimum score = 8 maximum score= 40) and lack of emotional awareness (minimum score = 5 maximum score = 25). the sub scales are summed to create the total score.

SECONDARY OUTCOMES:
Changes in the Acceptance and Action questionnaire II Questionnaire - II Acceptance and Action Questionnaire - II Acceptance and Action Questionnaire - II The acceptance and action questionnaire-II | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  The seven item questionnaire assesses psychological flexibility. Participants answer on a 1-7 likert scale, with higher scores indicating Higher scores indicating greater levels of psychological inflexibility. Minimum score = 7 and maximum score = 105.
Changes in the Brief symptom inventory | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  The brief symptom inventory is a 53 item self-report assessment designed to measure psychological distress as well as various psychological disorders/issues The BSI has nine subscales designed to assess individual symptom groups: somatization (SOM), obsessive-compulsive (OC), interpersonal sensitivity (IS), depression (DEP), anxiety (ANX), hostility (HOS), phobic anxiety (PHB, ), paranoid ideation (PAR), and psychoticism (PSY). The BSI also includes three scales that capture global psychological distress. Participants answer on a 0-4 likert scale, with higher scores indicating greater levels of psychopathology psychological issues. The minimum raw score is 0 and the maximum raw score is 212. Raw scores are converted to t-scores. The t-scores range from 30 to 80, with higher t-scores indicating greater disfunction. The global score equals the sum of all 53 items
Skills Use Follow-up questionnaire | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  This questionnaire asks participants if/how many times they have used the skills taught in the skills group since participating in the group. Responses range from 0 to 100, with higher numbers equating to higher usage of the skills.
Changes in the five facets of mindfulness questionnaire 15 item | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  This 15 item self-report question is designed to measure mindfulness. Participants answer on a 1-5 likert scale, with higher scores indicating greater levels of mindfulness. Minimum score = 15 and maximum score = 75. There are five sub scales: Observing (minimum score = 3 maximum score = 15); describing (minimum score = 3 maximum score = 15); acting with awareness (minimum score = 3 maximum score = 15); Non-judging (minimum score = 3 maximum score = 15); and non-reactivity (minimum score = 3 maximum score = 15). the sub scales are summed to create the total score.
Changes in the Post Traumatic Stress Disorder checklist for the DSM five civilian version | pre-test (before beginning the intervention), 2 days post-test (after intervention completion), 1 month (after the completion of the intervention) and 3 month (after the completion of the intervention). The data will be uploaded at the end of the study
  This 20 item self-report scale it is designed to capture symptoms of PTSD. Participants answer on a 0-4 likert scale, with higher scores indicating higher levels of PTSD symptomology. Minimum score = 0 and maximum score = 80.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine T Benuto, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Linehan, M. Cognitive-behavioral treatment of borderline personality disorder. New York, New York: Guilford press; 1993.
- [Background] 2. Linehan, M. M. Skills training manual for treating borderline personality disorder. New York, New York: Guilford Press; 1993.
- [Background] 3. Linehan, M. DBT® skills training manual. New York, New York: Guilford Publications; 2014.
- [Background] 4. Iverson, K.M., Shenk, C., & Fruzzetti, A. E. Dialectical behavior therapy for women victims of domestic abuse; a pilot study. Prof Psychol Res Pr. 2009;40(3); 242-248. Doi: 10.1037/a0013476
- [Background] 5. Ahrendt, A., Newlands, R., & Benuto, L. (2017, May). DBT for dv: New model, same positive outcomes. Poster session presented at the Nevada Psychological Association (NPA) 2017 Annual Conference, Las Vegas, NV.
- [Background] 6. Lee, J., & Fruzzetti, A. E. Evaluating a Brief Group Program for Women Victims of Intimate Partner Abuse. J Trauma Stress Disor Treat 2017; 6(3). doi: 10/4172/2324-8947.1000174
- [Background] Axelrod SR, Perepletchikova F, Holtzman K, Sinha R. Emotion regulation and substance use frequency in women with substance dependence and borderline personality disorder receiving dialectical behavior therapy. Am J Drug Alcohol Abuse. 2011 Jan;37(1):37-42. doi: 10.3109/00952990.2010.535582. Epub 2010 Nov 22. PMID 21091162
- [Background] 8. Alavi, K., Modarres, G. M., Amin, Y. S. A., & Salehi, F. J. Effectiveness of group dialectical behavior therapy (based on core mindfulness, distress tolerance and emotion regulationcomponents) on depressive symptoms in university students. The Quarterly Journal of Fundamentals of Mental Health. 2011; 13(2); 124-135.
- [Background] Linehan MM, Schmidt H 3rd, Dimeff LA, Craft JC, Kanter J, Comtois KA. Dialectical behavior therapy for patients with borderline personality disorder and drug-dependence. Am J Addict. 1999 Fall;8(4):279-92. doi: 10.1080/105504999305686. PMID 10598211
- [Background] Soeteman DI, Hakkaart-van Roijen L, Verheul R, Busschbach JJ. The economic burden of personality disorders in mental health care. J Clin Psychiatry. 2008 Feb;69(2):259-65. doi: 10.4088/jcp.v69n0212. PMID 18363454
- [Background] van Asselt AD, Dirksen CD, Arntz A, Severens JL. The cost of borderline personality disorder: societal cost of illness in BPD-patients. Eur Psychiatry. 2007 Sep;22(6):354-61. doi: 10.1016/j.eurpsy.2007.04.001. Epub 2007 Jun 4. PMID 17544636
- [Background] Clough BA, Casey LM. Technological adjuncts to increase adherence to therapy: a review. Clin Psychol Rev. 2011 Jul;31(5):697-710. doi: 10.1016/j.cpr.2011.03.006. Epub 2011 Mar 24. PMID 21497153
- [Background] Van Ameringen M, Turna J, Khalesi Z, Pullia K, Patterson B. There is an app for that! The current state of mobile applications (apps) for DSM-5 obsessive-compulsive disorder, posttraumatic stress disorder, anxiety and mood disorders. Depress Anxiety. 2017 Jun;34(6):526-539. doi: 10.1002/da.22657. Epub 2017 Jun 1. PMID 28569409
- [Background] 14. Rounsaville, B. J., Carroll, K. M., & Onken, L. S. Methodological diversity and theory in the stage model: Reply to Kazdin. Clinical Psychology Science and Practice, 2001; 8(2), 152-154. Doi: 10.1093/clipsy/8.2.152
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658